CLINICAL TRIAL: NCT05369897
Title: Benefits of a Virtual Reality Based Cognitive Intervention for Attention and Working Memory
Brief Title: VR for Improving Attention and Working Memory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Collaborators: National Center for Research and Development, Poland (Other); Senopi AG (Unknown)
Responsible Party: Principal Investigator, Jakub Kazmierski, Assoc. Prof. MD, PhD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RNN/222/21/KE
Record Dates: First submitted 2022-04-21; First posted 2022-05-11 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Virtual Reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be randomly assigned to either the experimental or the control group, and will be blind to the group assignment.
  The data gathered before and after the intervention will be sent to an external statistical analyst blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR training (Experimental): VR training for at least 10 minutes at least three days per week, resulting in a total of at least 36 sessions (at least ~12 hours of training in total) for each participant, spread across three months. Each session will focus on cognitive training.
  Interventions: Device: VR training
- VR activity (Sham Comparator): VR activity for at least 10 minutes at least three days per week, resulting in a total of at least 36 sessions (at least ~12 hours of training in total) for each participant, spread across three months, with 360º images and videos but without the interactive cognitive training.
  Interventions: Device: VR activity

INTERVENTIONS:
Device: VR training — The intervention group will receive cognitive training through VR headsets three times a week for 12 weeks. The intervention will be delivered in a virtual setting using images and music. The participants will be allowed to select the type of music and virtual environment during the intervention. The intervention will include four modules targeting attention and working memory through immersive VR.
  Arms: VR training
Device: VR activity — High-quality 360º images and videos from natural environments, such as a relaxing mountain environment. The participants in the control group will not receive cognitive training.
  Arms: VR activity

SUMMARY:
The main objective of the study is to investigate the effects of using a set of Virtual Reality (VR)-based Digital Therapeutics (DTx) apps to improve the cognitive abilities of healthy (high-functioning) seniors. For the purposes of the study, high-functioning seniors are defined as being over the age of 65 years, while maintaining their functional independence with regards to activities of daily living, including the ability to go on a long walk and the ability to interact with common modern technology (e.g. using a smartphone to send a message).

The study focuses on improving the quality of life of older healthy people by facilitating cognitive training through VR. Healthy people aged 65-85 will be eligible for the project. If the participants meet the inclusion criteria, they will be invited to participate in the study and be provided with detailed information about the research project. Based on sample size calculations, up to two hundred (200) older adults are intended to be included in the project. The participants will use specially designed VR systems and activities aimed at improving their cognitive abilities.

DETAILED DESCRIPTION:
The participants that meet inclusion criteria will be randomly assigned to the experimental group or the control group. The participants in the experimental group will receive a cognitive intervention focused on attention and working memory through virtual reality handsets. The intervention will be delivered at home and monitored by the research team via wifi. The participants will be required to perform the cognitive training at least 3 times a week for 12 weeks (36 training sessions). The participants in the control group will see high definition images through VR handsets without cognitive training.

The CNS-Vital Signs, a computerized neuropsychological battery, will be used to assess primary outcomes (Working Memory and Complex Attention), and will be administered to the participants before the intervention and after 36 training sessions. Differences in performance on primary and secondary outcomes will be analyzed with a Linear Mixed Model Analysis of Variance for longitudinal outcomes. Measures of anxiety and well-being will also be registered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or in a stable medical condition
* Undisturbed locomotion
* Do not require care or help from others in their everyday functioning
* Are able to go on long walks unassisted
* Are able to use common modern technology unassisted (e.g. using a smartphone to send a message)

Exclusion Criteria:

* Presence of neuropsychiatric disorders, including mild cognitive impairment (MCI) - Montreal Cognitive Assessment (MoCA) score <26 points
* Abuse or addiction to alcohol, drugs and tranquilizers
* Blurred vision that cannot be corrected with lenses or glasses that fit under the VR headset
* Auditory pathologies causing a significant decrease in hearing unaided
* High sensitivity to motion sickness
* Proneness to migraines
* Subject epileptic
* Subject vulnerable
* Subject obese or frail, as assessed based on their Body Mass Index (BMI)
* Subject considered by the study investigator to be an unsuitable candidate to participate in the study, due to other relevant reasons

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Working memory | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessed with the "Working Memory" domain from the CNS Vital Signs (CNSVS) computerized neuropsychological battery. The range of scores is from 0 to 38, with higher scores indicating better performance.
  A positive change after the intervention corresponds to an improvement in performace from baseline to follow-up.
Attention | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessed with the "Complex Attention" domain from the CNS Vital Signs (CNSVS) computerized neuropsychological battery. The range of scores is from 0 to 76, with higher scores indicating better performance.
  A positive change after the intervention corresponds to an improvement in performace from baseline to follow-up.

SECONDARY OUTCOMES:
Cognitive functioning | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessment of cognitive performance across a wide range of cognitive subdomains on the CNS Vital Signs (CNSVS) computerized battery (composite memory, verbal memory, visual memory, psychomotor speed, reaction time, cognitive flexibility, processing speed, executive function, simple attention, motor speed). The range of scores is from 0 to 40 (depending on the test), with higher scores indicating better performance.
  A positive change after the intervention corresponds to an improvement in performace from baseline to follow-up.
Standard grip strength measurement using a dynamometer | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessment of grip strength as a key frailty indicator. The range of scores is from 0 to 90, with higher scores indicating higher grip strength.
  A positive change after the intervention corresponds to an improvement in performace from baseline to follow-up.
The quality of life and the level of perceived well-being | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessment of the quality of life and the level of perceived well-being by using the World Health Organization 5 Well-Being Index. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
  A positive change after the intervention corresponds to an improvement in well-being from baseline to follow-up.
Severity of anxiety symptoms | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessment of the severity of anxiety symptoms by using Generalized Anxiety Disorder Questionnaire (GAD-7). The range of scores is from 0-21, with higher scores suggesting more severe ansiety symptoms.
  A positive change after the intervention corresponds to an increase in anxiety symptoms from baseline to follow-up.
Health-related quality of life | Change in scores between pre-intervention (baseline) and post-intervention (after 3 months).
  Assessment of the quantify the health-related quality of life by using the 5-level Euroquol 5D (EQ-5D-5L) questionnaire.
  The EQ-5D-5L questionnaire has 5 dimensions, each with 5 levels of perceived problems describing 3125 distinct health states: no problems (level 1), slight problems (level 2), moderate problems (level 3), severe problems (level 4), and extreme problems (level 5). EQ-5D-5L is a widely used measure of health-related quality of life.
  A positive change in the level of problems corresponds to an increase in the severity of symptoms from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Kaźmierski, PhD, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Department of Old Age Psychiatry and Psychotic Disorders Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
Once the first publication is publicly accessible, the anonymous data generated will be made available for sharing upon request. Shared data will include demographics, primary and secondary outcomes, and VR usability data. A committee of experts within the study team will discuss and decide whether data sharing is appropriate, based on the novelty and scientific rigor of the proposal. Applicants will be asked to sign a data access agreement to ensure a commitment to using the data only for research purposes and to securing the data with appropriate procedures. Redistribution of the data to other third parties will not be allowed.
Time Frame: Data will become available after the first publication. There is no time restriction for sharing the data.
Access Criteria: Through formal application. Applicants will be asked to sign a data access agreement to ensure a commitment to using the data only for research purposes and to securing the data with appropriate procedures.

REFERENCES:
- [Derived] Szczepocka E, Mokros L, Kazmierski J, Nowakowska K, Lucka A, Antoszczyk A, Oltra-Cucarella J, Werzowa W, Hellevik MM, Skouras S, Bagger K. The Effectiveness of Virtual Reality-Based Training on Cognitive, Social, and Physical Functioning in High-Functioning Older Adults (CoSoPhy FX): 2-Arm, Parallel-Group Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 5;13:e53261. doi: 10.2196/53261. PMID 38837194
- [Derived] Szczepocka E, Mokros L, Kazmierski J, Nowakowska K, Lucka A, Antoszczyk A, Oltra-Cucarella J, Werzowa W, Hellevik M, Skouras S, Bagger K. Virtual reality-based training may improve visual memory and some aspects of sustained attention among healthy older adults - preliminary results of a randomized controlled study. BMC Psychiatry. 2024 May 8;24(1):347. doi: 10.1186/s12888-024-05811-2. PMID 38720251